CLINICAL TRIAL: NCT06753721
Title: An Open-label, Multicenter, Single-arm Clinical Study on the Use of Doxorubicin Liposome in Combination With CapOX and Bevacizumab Regimen for First-line Treatment of Advanced Colorectal Adenocarcinoma With SMAD4R361H/C Mutation.
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2024-310
Record Dates: First submitted 2024-12-23; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Advanced Colorectal Adenocarcinoma
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Doxorubicin liposome combined with CapOX and Bevacizumab regimen as first-line treatment (Experimental): 6-month progression-free survival rate (6-month PFS rate) of Doxorubicin liposome combined with CapOX and Bevacizumab regimen as first-line treatment for advanced colorectal adenocarcinoma with SMAD4R361H/C mutation.
  Interventions: Drug: Doxorubicin liposome combined with CapOX and Bevacizumab

INTERVENTIONS:
Drug: Doxorubicin liposome combined with CapOX and Bevacizumab — Bevacizumab (7.5 mg/kg, IV, Day 1) + Oxaliplatin (130 mg/m², IV, Day 1) + Capecitabine (1000 mg/m², oral, twice daily, for 14 days) + Doxorubicin liposome (20 mg/m², IV, Day 1), repeated every 3 weeks.

SUMMARY:
This is a prospective, single-arm clinical study designed to evaluate the 6-month progression-free survival rate (6-month PFS rate) of Doxorubicin liposome combined with CapOX and Bevacizumab regimen as first-line treatment for advanced colorectal adenocarcinoma with SMAD4R361H/C mutation. The study plans to recruit 13 patients. After receiving 8 cycles of induction therapy, patients whose efficacy is evaluated as complete response (CR), partial response (PR), or stable disease (SD) (according to RECIST 1.1) will enter maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

1. The patient voluntarily participates in the study, signs the informed consent form, and demonstrates good compliance;
2. Age 18 years or older (inclusive), regardless of gender;
3. Histologically and/or cytologically confirmed unresectable colorectal adenocarcinoma;
4. For left-sided colon cancer or rectal cancer patients, must be non-RAS wild-type;
5. Non-dMMR/MSI-H;
6. SMAD4R361H/C mutation;
7. No prior history of systemic chemotherapy;
8. ECOG performance status of 0 or 1;
9. Hematological tests (within 14 days without blood transfusion): neutrophil absolute count ≥ 1.5 × 10⁹/L, platelet count ≥ 100 × 10⁹/L, hemoglobin ≥ 90 g/L;
10. Liver function tests (AST and ALT ≤ 3 × ULN, bilirubin ≤ 1.5 × ULN; if liver metastasis is present, AST and ALT ≤ 5 × ULN);
11. Renal function (serum creatinine ≤ 1.5 × ULN or creatinine clearance (CCr) ≥ 60 mL/min);
12. Both male and female subjects of reproductive age must use effective contraception.

Exclusion Criteria:

1. Patients with known contraindications to Doxorubicin liposome, Oxaliplatin, Capecitabine, or Bevacizumab;
2. Patients who have received radiotherapy or any anti-tumor treatments (chemotherapy, targeted therapy, immunotherapy, radiofrequency ablation, traditional Chinese medicine with anti-tumor indications, immunomodulators, or tumor embolization, etc.);
3. Patients who have had other malignancies within the past 5 years or have concurrent malignancies (except for cured skin basal cell carcinoma and carcinoma in situ of the cervix);
4. Patients who have experienced significant clinical bleeding symptoms, obvious bleeding tendency, or hemoptysis within 3 months prior to treatment, or who have had venous/thrombotic events such as cerebrovascular accidents (including transient ischemic attacks, intracerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism within the previous 6 months; or require long-term anticoagulation treatment with warfarin or heparin, or require long-term antiplatelet therapy (aspirin ≥300 mg/day or clopidogrel ≥75 mg/day);
5. Patients with active cardiovascular diseases within 6 months before treatment, including myocardial infarction, severe/uncontrolled angina. Echocardiography showing left ventricular ejection fraction <50%, or poorly controlled arrhythmia;
6. Known history of primary immunodeficiency virus infection;
7. Patients with active or uncontrolled severe infections;
8. Any other disease, clinically significant metabolic abnormalities, physical examination abnormalities, or laboratory test abnormalities, and based on the investigator's judgment, there is reasonable suspicion that the patient has a condition or disease that is unsuitable for the use of the study drug;
9. Any situation that, in the investigator's opinion, could pose a risk to the patient receiving study drug treatment, interfere with the assessment of the study drug's safety, or affect the interpretation of results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2024-12-31 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
6-month progression-free survival (PFS) | 3 years
  Defined as the time between the first occurrence of disease progression (PD) or death after the patient receives the study drug, whichever occurs first.

IPD SHARING:
Plan to Share IPD: No